CLINICAL TRIAL: NCT07244133
Title: Comparative Effects Of Powerball Using Static and Dynamic Surface on Upper Limb Endurance and Coordination in Children With Down Syndrome
Brief Title: Effects of Powerball in Children With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/Aymun Javed
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome
Keywords: Down Syndrome (DS); Powerball,; Upper extremity, Children
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial (RCT) will be conducted on 28 children aged 6-10 years, diagnosed with Down Syndrome with reduced upper extremity endurance and coordination..
  After screening participants will undergo 3 weeks power ball endurance training session, consisting of structured, repetitive and goal directed activities. Power ball training 3 sessions per week with the duration of 30 mins each session. Group A will receive different upper extremity activities with power ball on static surface while Group B will receive same activities with power ball on dynamic surface using a BOSU ball. The whole session followed by warm up and cool down sessions for 5 minutes each. Endurance will be assessed through ABIL-HAND kids tool. To access the coordination BOT-2 subsets test will be used.
  Data will be assessed using SPSS 27.0.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention will be power ball exercises on static surface (Experimental): Participants will undergo 3 weeks power ball endurance training session, consisting of structured, repetitive and goal directed activities. Power ball training 3 sessions per week with the duration of 30 mins each session. Group A will receive different upper extremity activities with power ball on static surface.The whole session followed by warm up and cool down sessions for 5 minutes each.Endurance will be assessed through ABIL-HAND kids tool. To access the coordination BOT-2 subsets test will be used.
  Data will be assessed using SPSS 27.0.
  Interventions: Other: Power ball with static surface
- The intervention will be powerball exercises on dynamic surface (Experimental): Participants will undergo 3 weeks power ball endurance training session, consisting of structured, repetitive and goal directed activities. Power ball training 3 sessions per week with the duration of 30 mins each session. Group B will receive different upper extremity activities with power ball on dynamic surface.The whole session followed by warm up and cool down sessions for 5 minutes each. Endurance will be assessed through ABIL-HAND kids tool. To access the coordination BOT-2 subsets test will be used.
  Data will be assessed using SPSS 27.0.
  Interventions: Other: Powerball with dynamic surface

INTERVENTIONS:
Other: Power ball with static surface — Participants will undergo 3 weeks power ball endurance training session, consisting of structured, repetitive and goal directed activities. Power ball training 3 sessions per week with the duration of 30 mins each session. Group A will receive different upper extremity activities with power ball on static surface. The whole session followed by warm up and cool down sessions for 5 minutes each.
  Arms: The intervention will be power ball exercises on static surface
Other: Powerball with dynamic surface — Participants will undergo 3 weeks power ball endurance training session, consisting of structured, repetitive and goal directed activities. Power ball training 3 sessions per week with the duration of 30 mins each session.Group B will receive same activities with power ball on dynamic surface using a BOSU ball. The whole session followed by warm up and cool down sessions for 5 minutes each.
  Arms: The intervention will be powerball exercises on dynamic surface

SUMMARY:
This randomised clinical trial investigates the effects of powerball using static and dynamic surface on upper limb Endurance and coordination in children with Down Syndrome. The study involves 28 children with Down Syndrome aged 6-10 years, will be randomly assigned one of the two groups for 3 week intervention period.

Power ball training 3 sessions per week with the duration of 30 mins each session. Group A will receive different upper extremity activities with power ball on static surface while Group B will receive same activities with power ball on dynamic surface using a BOSU ball. The whole session followed by warm up and cool down sessions for 5 minutes each. Endurance will be assessed through ABIL-HAND kids tool. To access the coordination BOT-2 subsets test will be used.

Data will be assessed using SPSS 27.0.

DETAILED DESCRIPTION:
This Randomized Clinical Trial (RCT) investigates the Comparative Effects of Powerball using static and dynamic surface on Upper Limb Endurance and Coordination in Children with Down Syndrome.This programme was designed to enhance the coordination and endurance in children with Down Syndrome.The efficacy of this programme was investigated through RCT. Data will be collected from special schools or rehabilitation centers. Data will be conducted on 28 children aged 6-10 years,diagnosed with Down Syndrome with reduced upper extremity endurance and coordination..

After screening participants will undergo 3 weeks power ball endurance training session, consisting of structured, repetitive and goal directed activities. Power ball training 3 sessions per week with the duration of 30 mins each session. Group A will receive different upper extremity activities with power ball on static surface while Group B will receive same activities with power ball on dynamic surface using a BOSU ball. The whole session followed by warm up and cool down sessions for 5 minutes each. Endurance will be assessed through ABIL-HAND kids tool. To access the coordination BOT-2 subsets test will be used.

Data will be assessed using SPSS 27.0.

ELIGIBILITY:
Inclusion Criteria:

* Children with Down Syndrome

  * Aged between 6-10 years
  * Both Genders
  * Ability to follow commands and instructions

Exclusion Criteria:

* Children with any orthopedic and neurological conditions associated with the syndrome • Children with any other Genetic disorder.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
ABIL-HAND | Baseline- 1st week and 3rd week
  ABIL-HAND Kids Tool is used for the assessment of upper extremity endurance. It's a parent-reported measure of a child's manual ability (unilateral and bilateral hand use) in everyday tasks. Parents rate each of 21 activities as Impossible / Difficult / Easy. The item difficulty increases with bimanual involvement. The responses are expressed in form of logits. 0.90 is the reliability with a validity of 0.77

SECONDARY OUTCOMES:
BOT-2 | Baseline- 1st week and 3rd week
  BOT-2 is a tool used for upper extremity coordination. This test is used to measures control and coordination of arm and hand movements. In this test visual and manual motor coordination (e.g., jumping, catching, throwing) will be assessed by performing different activities. The reliability of this tool is 0.86

CONTACTS AND LOCATIONS:
Overall Officials: AYMUN JAVED, MSPT, Principal Investigator — Ripha International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blazquez-Fernandez A, Lopez-Hazas-Jimenez G, Fernandez-Vazquez D, Navarro-Lopez V, Fernandez-Gonzalez P, Marcos-Anton S, Molina-Rueda F, Cano-de-la-Cuerda R. Effects of the powerball(R) system on muscle strength, coordination, fatigue, functionality and quality of life in people with multiple sclerosis. A randomized clinical trial. J Neuroeng Rehabil. 2024 Mar 2;21(1):33. doi: 10.1186/s12984-024-01325-w. PMID 38431591